CLINICAL TRIAL: NCT03760016
Title: Moderate-Intensity Exercise Versus High-Intensity Interval Training to Recover Walking Post-Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: University of Delaware (Other); University of Kansas Medical Center (Other); Children's Hospital Medical Center, Cincinnati (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Pierce Boyne, Associate Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-5325; R01HD093694 (NIH)
Record Dates: First submitted 2018-11-26; First posted 2018-11-30 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: Rehabilitation; Locomotion; Aerobic; Intensity; Dosing
MeSH Terms: conditions — Stroke | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate-Intensity Aerobic Training (Active Comparator)
  Interventions: Behavioral: Moderate-Intensity Aerobic Training
- High-Intensity Interval Training (Experimental)
  Interventions: Behavioral: High-Intensity Interval Training

INTERVENTIONS:
Behavioral: Moderate-Intensity Aerobic Training — Overground and treadmill walking with speed continuously adjusted to maintain a target heart rate of 40 +/- 5% heart rate reserve, progressing up to 55 +/- 5% heart rate reserve.
  Arms: Moderate-Intensity Aerobic Training
Behavioral: High-Intensity Interval Training — Overground and treadmill walking with 30 second bursts at maximum speed alternated with 30-60 second passive recovery periods. Intended to achieve a target average heart rate above 60% heart rate reserve.
  Arms: High-Intensity Interval Training

SUMMARY:
The objective of this study is to determine the optimal training intensity and the minimum training duration needed to maximize immediate improvements in walking capacity in chronic stroke. A single-blind, phase II, 3-site randomized controlled trial has been planned. Fifty persons >6 months post stroke will randomize to either moderate-intensity aerobic locomotor training or high-intensity interval locomotor training; each for 45 minutes, 3x/week for up to 36 total sessions over approximately 12 weeks. Clinical measures of walking function, aerobic fitness, daily walking activity and quality of life will be assessed at baseline (PRE) and after 4, 8 and 12 weeks of training (POST-4WK, POST-8WK, POST-12WK).

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-80 years at time of consenting
2. Single stroke for which participant sought treatment, 6 months to 5 years prior to consent date
3. Walking speed <1.0 m/s on the 10-meter walk test
4. Able to walk 10m over ground with assistive devices as needed and no continuous physical assistance from another person (guarding and intermittent assistance for loss of balance allowed)
5. Able to walk at least 3 minutes on the treadmill at ≥0.13m/s (0.3 mph)
6. Stable cardiovascular condition (AHA class B, allowing for aerobic capacity <6 metabolic equivalents)
7. Able to communicate with investigators, follow a 2-step command and correctly answer consent comprehension questions

Exclusion Criteria:

1. Exercise testing uninterpretable for ischemia or arrhythmia (e.g. resting ECG abnormality that makes exercise ECG uninterpretable for ischemia and no other clinical testing from the past year available to rule out)
2. Evidence of significant arrhythmia or myocardial ischemia on treadmill ECG graded exercise test in the absence of recent (past year) more definitive clinical testing (e.g. stress nuclear imaging) with negative result
3. Hospitalization for cardiac or pulmonary disease within past 3 months
4. Implanted pacemaker or defibrillator
5. Significant ataxia or neglect (score of 2 on NIH stroke scale item 7 or 11)
6. Severe lower limb spasticity (Ashworth >2)
7. Recent history (<3 months) of illicit drug or alcohol abuse or significant mental illness
8. Major post-stroke depression (Patient Health Questionnaire [PHQ-9] ≥ 10) in the absence of depression management by a health care provider
9. Currently participating in physical therapy or another interventional study
10. Recent botulinum toxin injection to the paretic lower limb (<3 months) or planning to have lower limb botulinum toxin injection in the next 4 months
11. Foot drop or lower limb joint instability without adequate stabilizing device, as assessed by a physical therapist
12. Clinically significant neurologic disorder other than stroke or unable to walk outside the home prior to stroke
13. Other significant medical condition likely to limit improvement or jeopardize safety as assessed by a physical therapist (e.g. joint contracture, gait limited by pain)
14. Pregnancy
15. Previous exposure to fast treadmill walking (>3 cumulative hours) during clinical or research therapy in the past year

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierce Boyne, DPT, PhD, Principal Investigator — University of Cincinnati
Locations (3):
- United States (3):
  - University of Delaware, Newark, Delaware
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
We deposited the final, de-identified dataset and data documentation into the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Data and Specimen Hub (DASH) archive (URL below)
Supporting Information: Study Protocol, SAP
Time Frame: Data are available now and should remain available indefinitely.
Access Criteria: Established by the repository
URL: https://dash.nichd.nih.gov/study/424597

REFERENCES:
- [Result] Boyne P, Billinger SA, Reisman DS, Awosika OO, Buckley S, Burson J, Carl D, DeLange M, Doren S, Earnest M, Gerson M, Henry M, Horning A, Khoury JC, Kissela BM, Laughlin A, McCartney K, McQuaid T, Miller A, Moores A, Palmer JA, Sucharew H, Thompson ED, Wagner E, Ward J, Wasik EP, Whitaker AA, Wright H, Dunning K. Optimal Intensity and Duration of Walking Rehabilitation in Patients With Chronic Stroke: A Randomized Clinical Trial. JAMA Neurol. 2023 Apr 1;80(4):342-351. doi: 10.1001/jamaneurol.2023.0033. PMID 36822187
- [Derived] Boyne P, Miller A, Schwab-Farrell SM, Sucharew H, Carl D, Billinger SA, Reisman DS. Training Parameters and Adaptations That Mediate Walking Capacity Gains from High-Intensity Gait Training Poststroke. Med Sci Sports Exerc. 2025 Jul 1;57(7):1285-1296. doi: 10.1249/MSS.0000000000003691. Epub 2025 Mar 3. PMID 40025665
- [Derived] Miller A, Reisman DS, Billinger SA, Dunning K, Doren S, Ward J, Wright H, Wagner E, Carl D, Gerson M, Awosika O, Khoury J, Kissela B, Boyne P. Moderate-intensity exercise versus high-intensity interval training to recover walking post-stroke: protocol for a randomized controlled trial. Trials. 2021 Jul 16;22(1):457. doi: 10.1186/s13063-021-05419-x. PMID 34271979
- Available data/document: Individual Participant Data Set: 424597 — https://dash.nichd.nih.gov/study/424597

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Started | 27 | 28
Completed 4-week Testing | 26 | 27
Completed 8-week Testing | 23 | 24
Completed | 19 | 23
Not Completed | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (9.9) | 61.5 (9.9) | 62.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 16 | 20 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 26 | 28 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 23 | 17 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 28 | 55
Stroke chronicity [Mean (Standard Deviation); unit: years] — Time interval from stroke onset to consent date
  years | 2.7 (1.4) | 2.2 (1.2) | 2.5 (1.3)
Self-selected gait speed [Mean (Standard Deviation); unit: meters/second] | 0.65 (0.29) | 0.62 (0.33) | 0.63 (0.31)
6-minute walk test distance [Mean (Standard Deviation); unit: meters] | 248 (136) | 230 (130) | 239 (132)

OUTCOME MEASURES:

1. Primary Outcome: Six-Minute Walk Test Distance
Description: Total distance walked in 6 minutes in meters
Time Frame: Change Six-Minute Walk Test Distance from Baseline to 4 Weeks
Population: Results are from an intent-to-treat analysis using a linear mixed effects model that included all available time points (Baseline, 4-week, 8-week and 12-week) for all randomized participants and estimated contrasts for change from baseline to each time point. Missing data were handled with the maximum likelihood method.
Measure: Least Squares Mean (95% Confidence Interval); unit: meters
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
meters | 27 [6 to 48] | 12 [-9 to 33]

2. Primary Outcome: Six-Minute Walk Test Distance
Description: Total distance walked in 6 minutes in meters
Time Frame: Change Six-Minute Walk Test Distance from Baseline to 8 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: meters
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
meters | 58 [39 to 76] | 29 [9 to 48]

3. Primary Outcome: Six-Minute Walk Test Distance
Description: Total distance walked in 6 minutes in meters
Time Frame: Change Six-Minute Walk Test Distance from Baseline to 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: meters
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
meters | 71 [49 to 94] | 27 [3 to 50]

4. Secondary Outcome: Comfortable Gait Speed
Description: From 10-meter walk test, in meters per second
Time Frame: Change from Baseline to 4 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: m/s
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
m/s | 0.11 [0.06 to 0.15] | 0.02 [-0.02 to 0.07]

5. Secondary Outcome: Comfortable Gait Speed
Description: From 10-meter walk test, in meters per second
Time Frame: Change from Baseline to 8 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: m/s
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
m/s | 0.14 [0.08 to 0.20] | 0.06 [0.00 to 0.12]

6. Secondary Outcome: Comfortable Gait Speed
Description: From 10-meter walk test, in meters per second
Time Frame: Change from Baseline to 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: m/s
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
m/s | 0.19 [0.13 to 0.25] | 0.06 [0.00 to 0.12]

7. Secondary Outcome: Fast Gait Speed
Description: From 10-meter walk test, in meters per second
Time Frame: Change from Baseline to 4 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: m/s
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
m/s | 0.22 [0.16 to 0.28] | 0.01 [-0.05 to 0.07]

8. Secondary Outcome: Fast Gait Speed
Description: From 10-meter walk test, in meters per second
Time Frame: Change from Baseline to 8 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: m/s
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
m/s | 0.24 [0.17 to 0.32] | 0.09 [0.01 to 0.17]

9. Secondary Outcome: Fast Gait Speed
Description: From 10-meter walk test, in meters per second
Time Frame: Change from Baseline to 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: m/s
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
m/s | 0.28 [0.19 to 0.37] | 0.09 [-0.01 to 0.18]

10. Secondary Outcome: Aerobic Fitness
Description: Oxygen consumption rate at ventilatory threshold during treadmill graded exercise test, in milliliters per kilogram body mass per minute
Time Frame: Change from Baseline to 4 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/kg/min
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
mL/kg/min | 1.3 [0.4 to 2.2] | 0.4 [-0.5 to 1.3]

11. Secondary Outcome: Aerobic Fitness
Description: as for outcome 10
Time Frame: Change from Baseline to 8 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/kg/min
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
mL/kg/min | 2.0 [0.7 to 3.3] | 1.7 [0.3 to 3.1]

12. Secondary Outcome: Aerobic Fitness
Description: as for outcome 10
Time Frame: Change from Baseline to 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/kg/min
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
mL/kg/min | 1.9 [0.4 to 3.4] | 1.4 [-0.2 to 3.0]

13. Secondary Outcome: PROMIS-Fatigue Scale
Description: The Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Scale is an 8-item self-report questionnaire about symptoms of fatigue. Each item is rated from 1-5, where higher scores indicate greater fatigue. A total raw score is calculated by summing the scores for each item. The raw score is then translated into a T-score based on normative data. The T-score is a standardized score with a mean of 50 and a standard deviation of 10 for the U.S. general population, so a T-score of 60 (for example) would represent one SD higher (worse) fatigue than the average American.
Time Frame: Change from Baseline to 4 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: T score
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
T score | -1.7 [-4.0 to 0.6] | 0.0 [-2.3 to 2.3]

14. Secondary Outcome: PROMIS-Fatigue Scale
Description: as for outcome 13
Time Frame: Change from Baseline to 8 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: T score
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
T score | -3.0 [-5.5 to -0.5] | 1.0 [-1.6 to 3.6]

15. Secondary Outcome: PROMIS-Fatigue Scale
Description: as for outcome 13
Time Frame: Change from Baseline to 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: T score
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
T score | -1.1 [-3.7 to 1.5] | -0.1 [-2.7 to 2.5]

16. Other Pre Specified Outcome: Exercise Capacity
Description: Time to exhaustion during treadmill graded exercise test, recorded in minutes
Time Frame: Change from Baseline to 4 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
minutes | 1.8 [1.1 to 2.4] | 0.6 [-0.1 to 1.2]

17. Other Pre Specified Outcome: Exercise Capacity
Description: Time to exhaustion during treadmill graded exercise test, recorded in minutes
Time Frame: Change from Baseline to 8 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
minutes | 2.5 [1.5 to 3.4] | 1.6 [0.6 to 2.5]

18. Other Pre Specified Outcome: Exercise Capacity
Description: Time to exhaustion during treadmill graded exercise test, recorded in minutes
Time Frame: Change from Baseline to 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
minutes | 3.3 [2.2 to 4.4] | 2.2 [1.1 to 3.4]

19. Other Pre Specified Outcome: Peak Oxygen Consumption Rate
Description: Peak oxygen consumption rate during treadmill graded exercise test, in milliliters per kilogram body mass per minute
Time Frame: Change from Baseline to 4 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/kg/min
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
mL/kg/min | 1.5 [0.5 to 2.5] | 0.2 [-0.8 to 1.2]

20. Other Pre Specified Outcome: Peak Oxygen Consumption Rate
Description: Peak oxygen consumption rate during treadmill graded exercise test, in milliliters per kilogram body mass per minute
Time Frame: Change from Baseline to 8 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/kg/min
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
mL/kg/min | 2.1 [0.8 to 3.5] | 1.5 [0.0 to 2.9]

21. Other Pre Specified Outcome: Peak Oxygen Consumption Rate
Description: Peak oxygen consumption rate during treadmill graded exercise test, in milliliters per kilogram body mass per minute
Time Frame: Change from Baseline to 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/kg/min
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
mL/kg/min | 2.5 [0.8 to 4.2] | 1.5 [-0.3 to 3.3]

22. Other Pre Specified Outcome: Metabolic Cost of Gait
Description: Oxygen consumption rate relative to speed during treadmill graded exercise test, in milliliters per kilogram body mass per meter
Time Frame: Change from Baseline to 4 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/kg/m
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
mL/kg/m | -0.08 [-0.13 to -0.03] | -0.05 [-0.10 to 0.00]

23. Other Pre Specified Outcome: Metabolic Cost of Gait
Description: as for outcome 22
Time Frame: Change from Baseline to 8 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/kg/m
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
mL/kg/m | -0.10 [-0.14 to -0.05] | -0.08 [-0.13 to -0.03]

24. Other Pre Specified Outcome: Metabolic Cost of Gait
Description: as for outcome 22
Time Frame: Change from Baseline to 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/kg/m
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
mL/kg/m | -0.12 [-0.17 to -0.06] | -0.11 [-0.17 to -0.06]

25. Other Pre Specified Outcome: EuroQol 5D-5L (EQ-5D-5L)
Description: A 5-item questionnaire about quality of life, including: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each item is scored from 1 to 5, where lower scores indicate greater quality of life. A total misery score was calculated by summing the scores for each item (min 5, max 25).
Time Frame: Change from Baseline to 4 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
score | -0.9 [-1.8 to -0.1] | -0.2 [-1.1 to 0.7]

26. Other Pre Specified Outcome: EuroQol 5D-5L (EQ-5D-5L)
Description: as for outcome 25
Time Frame: Change from Baseline to 8 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
score | -0.6 [-1.5 to 0.3] | -0.4 [-1.3 to 0.5]

27. Other Pre Specified Outcome: EuroQol 5D-5L (EQ-5D-5L)
Description: as for outcome 25
Time Frame: Change from Baseline to 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
score | -0.1 [-1.0 to 0.8] | -0.6 [-1.5 to 0.3]

28. Other Pre Specified Outcome: Activities-specific Balance Confidence Scale
Description: A 16-item questionnaire that asks participants to rate their balance confidence during everyday tasks, as a percentage from 0-100%, where higher scores indicate greater balance self-efficacy. A total score from 0-100 is calculated by averaging the scores for each item.
Time Frame: Change from Baseline to 4 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
score | -2.7 [-7.2 to 1.7] | -4.6 [-9.1 to -0.1]

29. Other Pre Specified Outcome: Activities-specific Balance Confidence Scale
Description: as for outcome 28
Time Frame: Change from Baseline to 8 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
score | 1.6 [-3.1 to 6.4] | -1.8 [-6.7 to 3.1]

30. Other Pre Specified Outcome: Activities-specific Balance Confidence Scale
Description: as for outcome 28
Time Frame: Change from Baseline to 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 27 | 28
score | 2.5 [-2.7 to 7.7] | 0.6 [-4.7 to 5.9]

31. Other Pre Specified Outcome: Daily Walking Activity
Description: Mean daily step count recorded with activity monitor, recorded as steps per day
Time Frame: Change from Baseline to 4 Weeks
Population: Results are from a modified intent-to-treat analysis using a linear mixed effects model that included all available time points (Baseline, 4-week, 8-week and 12-week) for all randomized participants and estimated contrasts for change from baseline to each time point. Four participants (2 in the HIT group and 2 in the MAT group) had to be excluded because they had no valid days of step data collected outside of study visits. Other missing data were handled with the maximum likelihood method.
Measure: Least Squares Mean (95% Confidence Interval); unit: steps/day
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 25 | 26
steps/day | -56 [-718 to 605] | -102 [-816 to 612]

32. Other Pre Specified Outcome: Daily Walking Activity
Description: Mean daily step count recorded with activity monitor, recorded as steps per day
Time Frame: Change from Baseline to 8 Weeks
Population: as for outcome 31
Measure: Least Squares Mean (95% Confidence Interval); unit: steps/day
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 25 | 26
steps/day | -299 [-1220 to 623] | 359 [-787 to 1505]

33. Other Pre Specified Outcome: Daily Walking Activity
Description: Mean daily step count recorded with activity monitor, recorded as steps per day
Time Frame: Change from Baseline to 12 Weeks
Population: as for outcome 31
Measure: Least Squares Mean (95% Confidence Interval); unit: steps/day
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
Number analyzed (Participants) | 25 | 26
steps/day | 65 [-1381 to 1512] | 267 [-1529 to 2062]

ADVERSE EVENTS:
Time Frame: Duration of participant enrollment post-randomization, which was approximately 4 months for participants who completed the study
Arm/Group | High-Intensity Interval Training | Moderate-Intensity Aerobic Training
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/27 | 3/28
Other Adverse Events (participants affected / at risk) | 13/27 | 10/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Intensity Interval Training (N=27) | Moderate-Intensity Aerobic Training (N=28)
seizure (Nervous system disorders) | 0 (0) | 1 (1) — seizure leading to temporary hospitalization, judged to be unrelated to study procedures
fall with fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — fall with hip fracture, judged to be unrelated to study procedures
delirium (Nervous system disorders) | 0 (0) | 1 (1) — delirium leading to temporary hospitalization, judged to be unrelated to study procedures
stroke (Nervous system disorders) | 1 (1) | 0 (0) — recurrent stroke, judged to be unrelated to study procedures
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High-Intensity Interval Training (N=27) | Moderate-Intensity Aerobic Training (N=28)
Pain/soreness (Musculoskeletal and connective tissue disorders) | 8 | 7 — Pain/soreness related to treatment
Fatigue (General disorders) | 2 | 2 — Fatigue related to treatment
Lightheadedness (General disorders) | 3 | 4 — lightheadedness related to treatment
Fall (General disorders) | 3 | 0 — Fall without injury related to treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT03760016/Prot_001.pdf
  • Statistical Analysis Plan (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/16/NCT03760016/SAP_000.pdf